CLINICAL TRIAL: NCT05771493
Title: The Spinopelvic Parameters, Body Mass Index and Waist Circumference in Patients With Chronic Non-specific Low Back Pain: an Observational Cross-sectional Correlation Study
Brief Title: The Spinopelvic Parameters, Body Mass Index and Waist Circumference in Patientd Chronic Non-specific Low Back Pain
Status: Completed | Type: Observational
Sponsor: AZ Nikolaas (Other)
Responsible Party: Principal Investigator, Erik Van de Kelft, M.D., PhD, Head of neursurgery, AZ Nikolaas
Other Study IDs: Vitaz Sint-Niklaas
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Low Back Pain
Keywords: Weight,; Body mass index; Pelvic index; Waist circumference
MeSH Terms: conditions — Low Back Pain; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measurement of baseline characteristics — Calculation of the correlation between BMI, WC and PI

SUMMARY:
This pilot study aims at styding the correlations between body mass index, waist circumference and the potential for positional adaptation of the pelvis to support overweight or obesity

DETAILED DESCRIPTION:
Record cards of patients presenting with non specific low back pain between January 1st 2020 and December 23rd 2022 were analysed.

All included patients had undergone a full spine X-ray allowing to calculate the pelvic index (PI). Weight status was described in 4 categories, in-line with the WHO definitions; Underweight (boddy mass index (BMI)) < 18.5 kg/m²; normal weight BMI 18.5 - 24.9 kg/m² , overweight BMI 25 - 29.9 kg/m², and obesity BMI ≥ 30 kg/m². To identify people with increased BMI-values and central (abdominal) fat distribution, we used the waist circumference (WC). The cut-off points of waist measurement that are used are 102 cm and 88 cm for men and women respectively. A high sacral slope (SS) means a greater the lumbar curvature, which results in a dynamic back. Due to the correlation between SS and PI, people with high PI values generally have higher values of SS. Therefore types 1 and 2 have a low-grade PI and types 3 and 4 have a high-grade PI Analysis of 272 patient records, shows that the mean PI is significantly different in the group with a low WC compared with the group with a high WC. BMI and WC show a significant correlation with PI

ELIGIBILITY:
Inclusion Criteria:

* presenting with non-specific low back pain
* having undergone full spine X-ray during the diagnostic proces

Exclusion Criteria:

* patients with missing data
* double entry of patients

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 272 patients; 51.8% male, 3.7% underweight; 28.7 % normal weight; 34.2% overweight and 33.5% obees. 50.4% has high WC. Mean PI 57.78
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Spinopelvic parameters and correlation with BMI and WC | January 1st 2020 - December 23, 2022
  Cross sectional study

CONTACTS AND LOCATIONS:
Locations (1):
- Vitaz, Sint-Niklaas, Belgium

IPD SHARING:
Plan to Share IPD: No
This is an analysis of patient record forms. Sharing the information would be against the privacy protection